CLINICAL TRIAL: NCT00535444
Title: Health and Faith Working Together to Control Blood Pressure
Brief Title: Health and Faith Working to Control Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #G06-08-103-02A
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: Hypertension; parish nurse
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Control (Active Comparator): assisted appointment with physician
  Interventions: Other: Parish nurse visit

INTERVENTIONS:
Other: Parish nurse visit — One visit with the parish nurse in 2 weeks

SUMMARY:
Faith community nursing programs have grown out of churches as a response to the inequity of healthcare delivery to uninsured and underinsured communities. These programs provide outreach to community members and extend their services beyond just the parishioners of the churches, reaching more uninsured people than traditional medical services. Although faith community nursing programs have been established throughout the United States, no evaluation of these programs has been done. QueensCare is taking the lead in measuring the effect of parish nurses on health outcomes. In this project we have one specific aim: to measure the effect of parish nurse visits on blood pressure control on community-dwelling hypertensive patients. Our study will involve recruiting hypertensive patients from parish nurse led health fairs and interviewing subjects at the time of recruitment. Patients will either be randomized to parish nurse visits or primary care physician appointments. We will have a 4-month follow-up period with a re-check of blood pressures and an exit interview of the patient. From this study, we hope to better understand if parish nurse visits improve blood pressure and medication compliance among hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* We will be including adults who are 18 years and older who have attended a health fair or screening event at one of QueensCare Health and Faith Partnership parish nurse sponsored church events in Los Angeles.
* Patients must be either English or Spanish speaking.
* Patients will be enrolled by blood pressure readings at the screening event. We will be using the JNC 71 criteria for diagnosing hypertension.
* Patients with blood pressures above 140/90 will be defined as hypertensive.
* Diagnosed and previously undiagnosed hypertensive patients will be included in the study.
* The patient must also be able to come to the follow-up appointment in 4 months.

Exclusion Criteria:

* Pregnant women will not be included in the study.
* Patients who do not speak English or Spanish will be excluded from the study since we do not have the capacity to translate all our materials into multiple languages.
* Those deemed by the research assistant to be incapable to give informed consent (due to intoxication, dementia, or other causes) will also be excluded from the study.
* Patients younger than 18 years old will be excluded from the study.
* Patients who have seen a parish nurse in her office hours in the past 6 months will be excluded from the study. We do not want patients who have an already established relationship with a parish nurse to be enrolled in the study with the chance of being randomized to the physician-only arm, which would interrupt the continuity of care the patient is receiving from the parish nurse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Drop of 12.5 mm Hg in systolic blood pressure | within 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Arshiya A Baig, MD/MPH, Principal Investigator — UCLA RWJ CSP